CLINICAL TRIAL: NCT01152710
Title: Capecitabine as Radiosensitising Agent in Neoadjuvant Treatment of Locally Advanced Resectable Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Prof.assist. Vaneja Velenik, MD, PhD, Institute of Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 139/03/06
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Resectable Rectal Cancer Clinical Stage II and III
Keywords: capecitabine; chemoradiation; rectal cancer; phase II study
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Capecitabine — Chemotherapy with capecitabine of 1650 mg/m2 daily dose will be administered orally, divided into two equal doses given 12 hours apart, during radiotherapy(45 Gy 1,8 Gy/fr), including weekends
  Other Names: Xeloda

SUMMARY:
A Phase II study aimed to evaluate the efficacy and toxicity of preoperative chemoradiotherapy with capecitabine in locally advanced resectable rectal cancer.

DETAILED DESCRIPTION:
Preoperative chemoradiation has become a standard part of treatment protocols in stage II and III rectal cancer. Compared to postoperative chemoradiotherapy, the advantage of preoperative application of chemotherapeutics and irradiation includes improved compliance, reduced toxicity and downstaging of the tumour in a substantial number of patients. The latter may enhance the rate of curative surgery, permit sphincter preservation in patients with low-sited tumours and have a positive impact on the quality of life of these patients. Orally administered capecitabine (Xeloda®, Hoffmann - La Roche Ltd, Basel, Switzerland) mimics the pharmacokinetics of continuous 5-FU infusion and makes chemoradiotherapy more patient-friendly. The mechanism of capecitabine activation, preferably in tumour cells, may further enhance its efficacy and tolerability, offering the potential for an enhanced therapeutic ratio.The aim of the present phase II study was to evaluate the efficacy and toxicity of preoperative chemoradiotherapy with capecitabine in patients with locally advanced rectal cancer. The primary endpoint of the study is a pathologically determined complete remission rate (pCR) of the disease locally and regionally. Secondly, the rate of sphincter preservation in low-sited tumours, overall downstaging rate,toxicity and survival parameters will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified adenocarcinoma of the rectum,
* resectable clinical stage II or III (IUCC TNM classification 2002);
* no prior radiotherapy and/or chemotherapy;
* World Health Organisation (WHO) performance status < 2;
* age at diagnosis of 18 or older;
* and adequate bone marrow, liver, renal and cardiac function (no history of ischemic heart disease).

Exclusion Criteria:

* A history of prior malignancy other than non-melanoma skin cancer or in situ carcinoma of the cervix

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
complete pathological remission rate | 9 weeks
  after pathological examination of resected specimen

SECONDARY OUTCOMES:
the rate of sphincter preservation in low-sited tumours | 9 weeks
  after the operation
toxicity of combined modality treatment (Number of Participants with Adverse Events) | 5 weeks
  During preoperative treatment, patients will be evaluated weekly for acute toxicity and compliance with the protocol. Clinical examination and complete blood count will be performed and body weight was measured. Toxic side effects will be assessed according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) (version 2.0). Patients will be followed every three month for the first two years after the last cycle of adjuvant chemotherapy and thereafter every six month up to 5th year.
overall downstaging rate | 9 weeks
  after the pathological examination of resected specimen
overall survival | 5 years
  Overall survival is defined as the time from inclusion to the date of death from any cause or to the date of last follow-up.
local control | 5 years
  Local control is defined as the time from inclusion to the date of local recurrence
relapse-free survival | 5 years
  Relapse-free survival iss defined as the time from inclusion to the first occurrence of disease relapse (local or distant), death or date of last follow-up.
long-term rectal and urogenital morbidity | 2 years after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology, Ljubljana, Slovenia, Slovenia

REFERENCES:
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Schuller J, Cassidy J, Dumont E, Roos B, Durston S, Banken L, Utoh M, Mori K, Weidekamm E, Reigner B. Preferential activation of capecitabine in tumor following oral administration to colorectal cancer patients. Cancer Chemother Pharmacol. 2000;45(4):291-7. doi: 10.1007/s002800050043. PMID 10755317
- [Background] Kim JS, Kim JS, Cho MJ, Song KS, Yoon WH. Preoperative chemoradiation using oral capecitabine in locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2002 Oct 1;54(2):403-8. doi: 10.1016/s0360-3016(02)02856-0. PMID 12243814
- [Background] Twelves C, Boyer M, Findlay M, Cassidy J, Weitzel C, Barker C, Osterwalder B, Jamieson C, Hieke K; Xeloda Colorectal Cancer Study Group. Capecitabine (Xeloda) improves medical resource use compared with 5-fluorouracil plus leucovorin in a phase III trial conducted in patients with advanced colorectal carcinoma. Eur J Cancer. 2001 Mar;37(5):597-604. doi: 10.1016/s0959-8049(00)00444-5. PMID 11290435
- [Background] Jansman FG, Postma MJ, van Hartskamp D, Willemse PH, Brouwers JR. Cost-benefit analysis of capecitabine versus 5-fluorouracil/leucovorin in the treatment of colorectal cancer in the Netherlands. Clin Ther. 2004 Apr;26(4):579-89. doi: 10.1016/s0149-2918(04)90060-4. PMID 15189755
- [Background] Dunst J, Reese T, Sutter T, Zuhlke H, Hinke A, Kolling-Schlebusch K, Frings S. Phase I trial evaluating the concurrent combination of radiotherapy and capecitabine in rectal cancer. J Clin Oncol. 2002 Oct 1;20(19):3983-91. doi: 10.1200/JCO.2002.02.049. PMID 12351595
- [Result] Velenik V, Anderluh F, Oblak I, Strojan P, Zakotnik B. Capecitabine as a radiosensitizing agent in neoadjuvant treatment of locally advanced resectable rectal cancer: prospective phase II trial. Croat Med J. 2006 Oct;47(5):693-700. PMID 17042060